CLINICAL TRIAL: NCT02342951
Title: Evaluation of Lung Clearance Index for Early Detection of Lung Disease in Young Children With Cystic Fibrosis
Brief Title: Evaluation of the Lung Clearance Index
Acronym: LCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Vaincre la Mucoviscidose (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: RCB-2013-A01175-40
Record Dates: First submitted 2014-08-07; First posted 2015-01-21 (Estimated); Last update posted 2019-10-21 (Actual); Status verified 2019-10

CONDITIONS: Cystic Fibrosis
Keywords: Cystic fibrosis,; lung clearance index,; pulmonary function
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LCI (Other): Measure of lung clearance index
  Interventions: Other: Lung clearance index determination

INTERVENTIONS:
Other: Lung clearance index determination — Lung clearance index determination

SUMMARY:
The purpose of this study is to determine the efficacy of a non invasive method of detecting the pulmonary disease in order to initiate treatment against cystic fibrosis as soon as possible.

Moreover this screening procedure permits to note the improvement following the treatment and to choose the optimal treatment in term of efficacy.

DETAILED DESCRIPTION:
It is mandatory to detect as early as possible lung CF disease in the young child with CF to initiate active therapies limiting irreversible lesions. Lung Clearance Index (LCI) which evaluates gas clearance from the alveolar volume is an easy to-do technique in pre-school children.

Main objective To evaluate correlation between LCI and thoracic low dose computed tomodensitometry (CT) endpoints at initial visit Secondary objectives

1. To evaluate correlation between LCI and respiratory function measurements at each visit
2. To evaluate correlation between the evolution of LCI and respiratory function endpoints and the evolution of CT only for the children for whom a thoracic low dose CT is requested by their referent doctor after two years.
3. To evaluate LCI predictive value for respiratory function 2 years later in preschool children.

This is a prospective multicenter cohort study. Study visits will be performed each year during the annual check up for normal follow up of the child.

Initial visit (Visit 1) takes place during an annual check-up during which a low dose CT was prescribed. It will include following tests: LCI, Lung function tests (LFTs) performed according to age (forced volumes and flows, plethysmographic specific airway resistances and interrupter resistances), and a low dose CT scan performed according a standardized protocol.

Visit 2 will be performed 12 ± 3 months later and will include following tests: LCI , LFTs.

Visit 3 will be performed 24 ± 3 months later and will include following tests: LCI , LFTs and, if judged necessary by the child's referent doctor, a low dose CT scan performed according to a standardized protocol.

Anthropometric data, infection history, treatment will be collected at each visit.

Recruiting period: 1 year Study period: 2 years per patient, 3 years as a whole LCI will help to evaluate early ventilation inhomogeneity due to small bronchi abnormalities in young children with CF. Concordance between LCI and CT endpoints evaluation will help to define the frequency of lung CT administration in young CF children. Predictive value for later abnormal lung function development will be evaluated. This will help to detect the children at risk to develop abnormal lung function and to target those requiring active treatment. Finally this endpoint will be very valuable in the future therapeutic trials for CFTR correctors or potentiators.

ELIGIBILITY:
Inclusion Criteria:

* Children with typical cystic fibrosis (sweat chloride level >60 mEq/l) followed in reference centre participating to the study
* From 3 to 6 years old
* Children with a planned annual assessment that required thoracic computed tomography and lung function test
* Children with informed and non opposed parents

Exclusion Criteria:

* Children with atypical cystic fibrosis
* Children with bronchial exacerbation dating less than 2 weeks
* Children with severe associated disease

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 53 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2019-04 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
measure of nitrogen washout and Brody 2 score | Month 0

SECONDARY OUTCOMES:
measure of FEV (Correlation between the evolution of LCI and respiratory function endpoints and CT) | 2 years
  Correlation between the evolution of LCI and respiratory function endpoints and CT
measure of FEV (Evaluation of LCI predictive value for respiratory function in preschool children) | 2 years
  Evaluation of LCI predictive value for respiratory function in preschool children.

CONTACTS AND LOCATIONS:
Overall Officials: Muriel Le Bourgeois, MD, Principal Investigator — Service de pneumologie pédiatrique, Hôpital Necker-Enfants Malades Assistance Publique Hôpitaux de Paris 75015 Paris, France
Locations (1):
- Hôpital Necker-Enfants Malades, Paris, France